CLINICAL TRIAL: NCT05830877
Title: The RCT Study on the Evaluation of Clinical Effect of Primary Insomnia Treated With the Tiaoshen Acupuncture
Brief Title: The Study on the Evaluation of Acupuncture Therapy on Primary Insomnia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Liu Yingjun, Attending doctor, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023ZL476
Record Dates: First submitted 2023-04-01; First posted 2023-04-26 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Primary Insomnia
Keywords: acupuncture; Primary Insomnia; RCT
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the acupuncture group (Experimental): the patients included in this arm will recept the Tiaoshen acupuncture.
  Interventions: Other: the acupuncture group
- the placebo acupuncture group (Active Comparator): Subjects in the placebo acupuncture group will receive non-insertive acupuncture using the sham needle supported by the Park device, and the selected acupoints is the same as the acupuncture group.
  Interventions: Other: the placebo acupuncture group

INTERVENTIONS:
Other: the acupuncture group — The primary choice is to puncture GB20 with a quick puncture, which means "regulate the mind and open the way". ①Scalp acupuncture: Du 20(Baihui), EX-HN 3(Yintang), EX-HNl(Sishencong); ②Select acupoints from six acupoints for mind-regulating, ear points (both sides): heart, lung, and Shenmen; body points (both sides): LI20(Yingxiang), EXTRA 12(Anmian), ST36(Zusanli) as the main hole. ③Sleeping three needles(both sides): HT7(Shenmen), PC6(Neiguan), SP6(Sanyinjiao); ④Opening four gates: LI4(Hegu) , LR3(Taichong) ⑤Abdominal four needles:ST25(Tianshu), CV12(Zhongwan), CV4(Guanyuan). For body acupuncture, a 0.3 mm×40 mm needle was used to insert directly for 0.5-1.0 cun, and twisting to gain the qi; for auricular points, a 0.25 mm×40 mm needle was used for 2-3 minutes without manipulating the needle. The acupuncture points were retained for 30 min, and the treatment was performed once every other day, three times a week, and the curative effect was evaluated after 4 weeks of treatment.
  Arms: the acupuncture group
Other: the placebo acupuncture group — Subjects in the placebo acupuncture group will receive non-insertive acupuncture using the sham needle supported by the Park device. This needle has a retractable shaft and a blunt tip, they could not penetrate the skin. We gently placed the sham needle and Park device on the skin. The sham needle is then no longer manipulated to minimize any physiological effects. The selected acupoints and needle retention time were the same as for the acupuncture group. Since oblique insertion is required for acupuncture points on the head, the fixed acupuncture body of the Park device could not be used. Therefore, blunt needles are used to stimulate the head points to reduce the amount of stimulation produced by acupuncture. At the end of the treatment, the acupuncturist also used a dry cotton swab to press the acupoints so that patients could feel the withdrawal of 'real' needles.
  Arms: the placebo acupuncture group

SUMMARY:
Through the recruition of outpatients who clinically meet the diagnostic criteria and inclusion criteria of PI, the acupuncture group adopts Tiaoshen acupuncture, and the placebo acupuncture group adopts non-insertive acupuncture supported by the Park device, and the Pittsburgh Sleep Quality Index (PSQI) is used as the main index to evaluate the patients through the scale; subjective indicators like Chalder 14-item fatigue scale, Epworth sleepiness rating, self-rating anxiety scale (SAS), self-rating depression scale (SDS) and objective indicators like polysomnography (PSG), heart rate variability (HRV) is regarded as a secondary index, and then evaluate the clinical efficacy of Tiaoshen acupuncture on PI and explore its mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Conforming to the diagnostic criteria of traditional Chinese and Western medicine for chronic insomnia;
* Age range: 18-70 years old;
* PSQI score>7 points; SAS score > 50 or SDS score > 53;
* No communication and cognitive impairment;
* No use or withdrawal of psychoactive drugs such as anti-anxiety within one month; ·No major physical diseases;
* Those who voluntarily accept the research content and can complete various scale evaluations, polysomnography monitoring and HRV;
* Sign an informed consent form prior to the start of the study.

Exclusion Criteria:

* Those who do not meet the inclusion criteria;
* Persons with a history of severe mental illness, severe head injury, and significant disturbance of consciousness;
* Those with severe liver and renal insufficiency and bleeding tendencies;
* Alcoholism (liquor ≥ 100ml/day), smoking (≥ 15 cigarettes/day), drug abuse or taking psychotropic drugs;
* People with other sleep disorders, such as sleep apnea hypopnea syndrome, paroxysmal sleeping sickness, and REM sleep behavioral disorders;
* Pregnant or nursing;
* Those with other major diseases and poor control;
* Other persons who are unwilling to sign informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh sleep quality index | Before treatment
  Use the PSQI score table to evaluate according to patient's situation, and analyze the score changes of the subjects' insomnia degree before and after treatment by the analysis of score data. The PSQI consists of 19 self-rated questions and 5 questions rated by sleep partners. The 19 self-assessment questions constitute 7 factors ranging from 0 to 3 points. The cumulative score of each factor component is the total score of the PSQI, and the total score ranges from 0 to 21. The higher the score, the worse the sleep quality.
Pittsburgh sleep quality index | the 4th week of treatment
  Use the PSQI score table to evaluate according to patient's situation, and analyze the score changes of the subjects' insomnia degree before and after treatment by the analysis of score data. The PSQI consists of 19 self-rated questions and 5 questions rated by sleep partners. The 19 self-assessment questions constitute 7 factors ranging from 0 to 3 points. The cumulative score of each factor component is the total score of the PSQI, and the total score ranges from 0 to 21. The higher the score, the worse the sleep quality.
Pittsburgh sleep quality index | 4 weeks after treatment
  Use the PSQI score table to evaluate according to patient's situation, and analyze the score changes of the subjects' insomnia degree before and after treatment by the analysis of score data.The PSQI consists of 19 self-rated questions and 5 questions rated by sleep partners. The 19 self-assessment questions constitute 7 factors ranging from 0 to 3 points. The cumulative score of each factor component is the total score of the PSQI, and the total score ranges from 0 to 21. The higher the score, the worse the sleep quality.

SECONDARY OUTCOMES:
Fatigue Scale-14 | Before treatment
  Respond to the severity of fatigue from different angles through 14 questions.The Fatigue Scale-14 is composed of 14 items, and the 14 items are divided into two categories. One category reflects physical fatigue, including 1 to 8 items; the other reflects mental fatigue, including 9 to 14 in total 6 items. The highest score for physical fatigue is 8, the highest score for mental fatigue is 6, and the highest total score is 14. The higher the score, the more severe the fatigue.
Fatigue Scale-14 | the 4th week of treatment
  Respond to the severity of fatigue from different angles through 14 questions.The Fatigue Scale-14 is composed of 14 items, and the 14 items are divided into two categories. One category reflects physical fatigue, including 1 to 8 items; the other reflects mental fatigue, including 9 to 14 in total 6 items. The highest score for physical fatigue is 8, the highest score for mental fatigue is 6, and the highest total score is 14. The higher the score, the more severe the fatigue.
Fatigue Scale-14 | 4 weeks after treatment
  Respond to the severity of fatigue from different angles through 14 questions.The Fatigue Scale-14 is composed of 14 items, and the 14 items are divided into two categories. One category reflects physical fatigue, including 1 to 8 items; the other reflects mental fatigue, including 9 to 14 in total 6 items. The highest score for physical fatigue is 8, the highest score for mental fatigue is 6, and the highest total score is 14. The higher the score, the more severe the fatigue.
Epworth Sleepiness Scale | Before treatment
  The epworth sleepiness scale is applied to assess excessive daytime sleepiness. The clinical significance of this table is: sleepiness can be semi-objectively assessed by the epworth sleepiness scale. Any sleep disorder caused by sleep deprivation may lead to change of this scale. This scale has 24 points. A score greater than 6 indicates drowsiness, a score greater than 11 indicates excessive sleepiness, and a score greater than 16 indicates dangerous drowsiness.
Epworth Sleepiness Scale | he 4th week of treatment
  The epworth sleepiness scale is applied to assess excessive daytime sleepiness. The clinical significance of this table is: sleepiness can be semi-objectively assessed by the epworth sleepiness scale. Any sleep disorder caused by sleep deprivation may lead to change of this scale. This scale has 24 points. A score greater than 6 indicates drowsiness, a score greater than 11 indicates excessive sleepiness, and a score greater than 16 indicates dangerous drowsiness.
Epworth Sleepiness Scale | 4 weeks after treatment
  The epworth sleepiness scale is applied to assess excessive daytime sleepiness. The clinical significance of this table is: sleepiness can be semi-objectively assessed by the epworth sleepiness scale. Any sleep disorder caused by sleep deprivation may lead to change of this scale. This scale has 24 points. A score greater than 6 indicates drowsiness, a score greater than 11 indicates excessive sleepiness, and a score greater than 16 indicates dangerous drowsiness.
Self-Rating Anxiety Scale | Before treatment
  SAS is called anxiety self-rating scale, which is a standard for anxiety assessment and a psychological scale used to measure the degree of anxiety state and its changes during treatment. The SAS scale has 100 points in total, and the cut-off value is 50 points, of which 50-59 points are mild anxiety, 60-69 points are moderate anxiety, and more than 70 points are severe anxiety.
Self-Rating Anxiety Scale | 4th week of treatment
  SAS is called anxiety self-rating scale, which is a standard for anxiety assessment and a psychological scale used to measure the degree of anxiety state and its changes during treatment. The SAS scale has 100 points in total, and the cut-off value is 50 points, of which 50-59 points are mild anxiety, 60-69 points are moderate anxiety, and more than 70 points are severe anxiety.
Self-Rating Anxiety Scale | 4 weeks after treatment
  SAS is called anxiety self-rating scale, which is a standard for anxiety assessment and a psychological scale used to measure the degree of anxiety state and its changes during treatment. The SAS scale has 100 points in total, and the cut-off value is 50 points, of which 50-59 points are mild anxiety, 60-69 points are moderate anxiety, and more than 70 points are severe anxiety.
Self-rating depression scale | Before treatment
  The depression self-rating scale is a standard for depression assessment, which can quite intuitively reflect the subjective feelings of depressed patients during treatment. It is mainly applicable to adults with depressive symptoms, including outpatients and inpatients. The SDS scale has 100 points in total, and the cut-off value is 53 points, of which 53-62 points are mild anxiety, 63-72 points are moderate anxiety, and more than 73 points are severe anxiety.
Self-rating depression scale | the 4th week of treatment
  The depression self-rating scale is a standard for depression assessment, which can quite intuitively reflect the subjective feelings of depressed patients during treatment. It is mainly applicable to adults with depressive symptoms, including outpatients and inpatients. The SDS scale has 100 points in total, and the cut-off value is 53 points, of which 53-62 points are mild anxiety, 63-72 points are moderate anxiety, and more than 73 points are severe anxiety.
Self-rating depression scale | 4 weeks after treatment
  The depression self-rating scale is a standard for depression assessment, which can quite intuitively reflect the subjective feelings of depressed patients during treatment. It is mainly applicable to adults with depressive symptoms, including outpatients and inpatients. The SDS scale has 100 points in total, and the cut-off value is 53 points, of which 53-62 points are mild anxiety, 63-72 points are moderate anxiety, and more than 73 points are severe anxiety.
Polysomnography | the 4th week of treatment
  Polysomnography refers to the continuous and synchronous acquisition, recording and analysis of EEG, electrooculogram, electromyogram, oronasal airflow, respiratory effort, and saturation of oxygen levels, body position and other physiological and pathological parameters during sleep by sleep technicians all night through computer software in the sleep laboratory. This technology for the diagnosis of sleep disorders is the gold standard for the diagnosis and treatment of sleep disorders.
Heart rate variability | the 4th week of treatment
  Heart rate variability (HRV) refers to the fluctuations in the interval between successive heartbeats. It is commonly used to evaluate the regulatory role of the autonomic nervous system on cardiac activity. It is an important noninvasive indicator for evaluating autonomic nervous activity, and is also one of the important indicators for evaluating autonomic nervous changes during sleep.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China